CLINICAL TRIAL: NCT00682175
Title: Metabolic Derangements in Acute Heart Failure Syndrome
Status: Terminated | Type: Observational
Why Stopped: Project not initiated
Sponsor: The Cleveland Clinic (Other)
Responsible Party: George Sokos, MD, Cleveland Clinic Foundation
Other Study IDs: 08-169
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Adult (age > 18 yrs) patients admitted to the Heart Failure Intensive Care Unit with Acute Heart Failure Syndrome requiring placement of a Pulmonary Artery catheter for hemodynamically guided therapy.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Pulmonary Artery pressure (PA), pulmonary capillary wedge pressure (PCWP), cardiac output (CO), and cardiac index (CI). This data will be collected after 24 ± 2 and 48 ± 2 hours of standard heart failure therapy

SUMMARY:
To determine the association of both neurohormonal and hemodynamic alterations associated with metabolic abnormalities in acute heart failure syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 yrs) patients admitted to the Heart Failure Intensive Care Unit (H22) with Acute Heart Failure Syndrome (AHFS) requiring placement of a Pulmonary Artery catheter for hemodynamically guided therapy.

Exclusion Criteria:

* History of Congenital Heart Disease.
* Acute HF in the setting of acute myocardial infarction.
* Severe Anemia
* Patients listed for cardiac transplantation.
* Terminal Malignancy, AIDS or CNS disease.
* Concomitant sepsis, ARDS, trauma, aortic dissection, or pericardial tamponade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age > 18 yrs) patients admitted to the Heart Failure Intensive Care Unit (H22) with Acute Heart Failure Syndrome (AHFS) requiring placement of a Pulmonary Artery catheter for hemodynamically guided therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Sokos, MD, Principal Investigator — The Cleveland Clinic